CLINICAL TRIAL: NCT06198855
Title: Automated Measurement of Blood Pressure in Waiting Appointment Versus 24-h Ambulatory Measurements
Brief Title: Automated Measurement of Blood Pressure in Waiting Room (AMBP-waiting)
Acronym: AMBP-waiting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación para la Formación e Investigación de los Profesionales de la Salud de Extremadura (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Other Study IDs: DTS19/00003
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-12

CONDITIONS: Blood Pressure; Hypertension; Blood Pressure Measurement
Keywords: Blood Pressure measurement.; Automatic Blood Pressure office assessment.
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertension Diagnosis: Subject need 24-h BP monitor for hypertension diagnosis
  Interventions: Device: QMon-20 device
- hypertension control evaluation: Patients need 24-h BP monitor for assessment hypertension control
  Interventions: Device: QMon-20 device

INTERVENTIONS:
Device: QMon-20 device — Automatic Blood pressure measurement with QMon-20 device in the waiting room for 20 minutes every 5 minutes.
  Other Names: 24-h monitor BP

SUMMARY:
The investigators will study 500 patients with any indication for 24-hours Ambulatory Blood Pressure Monitoring (ABPM). In this study will compare Blood Pressure measurements with an original automatic device every 5 minutes during 20 minutes while the subject waits room for appointment, against ABPM results.

DETAILED DESCRIPTION:
The objective in the care of the hypertensive patient must be to establish a correct diagnosis and obtain a correct control of the BP, with the ultimate aim of reducing cardiovascular morbidity and mortality. Classically, a degree of knowledge of 50% of the hypertensive population has been considered; 50% of these received treatment, and 50% of the latter were controlled, which means a control of 25% of known hypertensive patients. The causes that lead to this deficit control are varied: Low degree of treatment completion, therapeutic inertia - static therapeutic attitude to the poorly controlled patient - and the incorrect measurement of blood pressure values. Therefore, within the control measures to control hypertension, an effort should be made to improve blood pressure measurement techniques. Accurate knowledge of blood pressure (BP) figures is critical for diagnosis, prognosis and therapeutic decision. However, despite the magnitude of the problem and the huge amount of clinical studies, physicians continue to need an optimal technique that can be applied in daily practice. Even in the main population-based studies, such as NHANES, they compared the control of BP with different measurement methods. More recently, the method applied in the SPRINT study has raised great controversy. This technique consists in the measurement of automatic BP in office without the presence of health personnel(ABPM-office), largely avoiding the white coat effect. Their results have influenced the change in the diagnostic figures of hypertension and therapeutic objectives in the recommendations of the American and European guidelines.

This new method was recommended by some scientific societies and in the future could become a reference technique for measuring BP in appointment. A has been shown to obtain readings similar to those of 24h-ABPM and its clinical utility has been demonstrated in a large randomized clinical trial, CAMBO. This method was used in the SPRINT study and some scientific societies have proposed it for the diagnosis of hypertension and recommending it if we do not have 24h-ABPM or it is necessary to perform repeated assessments of BP. The Canadian Society of Hypertension has officially recommended its use and the technique is regularly used by more than 50% of primary care physicians. Despite the positive results, both in US and Europe, this technique has drawbacks that limit its generalization in real-life. The setting of commercial devices are limited and their are compact, table-top device that does not allow patient mobilization. Finally, examination should be performed with the patient alone, in a quiet place and close to the consultation that is rarely available in many health systems.

Therefore,availability of an easy-to-use, portable BP device, which allows BP measured automatically while the patient waits in the medical consultation room, could avoid the white coat effect by providing a accurate BP measurement and avoid a large number of studies.

ELIGIBILITY:
Inclusion Criteria:

* Indication for 24-h holter pressure study for hypertension diagnosis.
* Indication for 24-h holter pressure study for assess hypertension control

Exclusion Criteria:

* Any inability to perform 24-h ambulatory BP measurements.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Patients with clinical indication to perform 24-h BP measurement study due to hypertension diagnostic
  Group 2: Patients with clinical indication to perform 24-h BP measurement study due to hypertension control
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
concordance of systolic and diastolic BP mean between waiting room measurements and 24-h monitor mean. | 6 MONTHS
  mm Hg differences between measurements in the office with 24-h monitor
concordance of systolic and diastolic BP mean between waiting room measurements and 24-h diurnal monitor mean. | 6 MONTHS
  mm Hg differences between measurements in the office with 24-h monitor

CONTACTS AND LOCATIONS:
Overall Officials: JUAN F SANCHEZ M-TORRERO, PhD, Principal Investigator — Universidad Extremadura

IPD SHARING:
Plan to Share IPD: Yes
Recruitment in others hospital.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months

REFERENCES:
- [Result] Robles NR, Sanchez Munoz-Torrero JF. Automated blood pressure measurement in consultation. Med Clin (Barc). 2020 Jan 24;154(2):59-60. doi: 10.1016/j.medcli.2019.04.009. Epub 2019 Jun 11. No abstract available. English, Spanish. PMID 31196667
- [Result] Rico-Martin S, Sanchez-Bacaicoa M, Calderon-Garcia JF, Labrador-Gomez PJ, De Nicolas Jimenez JM, Villa-Rincon J, Robles NR, Guijarro C, Iammarino C, Rodilla-Salas E, Sanchez Munoz-Torrero JF. Validation of the QMon-20 oscillometric blood pressure monitor for professional office use in the general population according to the ANSI/ESH/ISO 81060-2:2018 protocol. Blood Press Monit. 2021 Oct 1;26(5):393-395. doi: 10.1097/MBP.0000000000000540. PMID 34001760
- [Derived] Sanchez Bacaicoa M, Rico S, Gullon A, Fernandez Pardo J, Villa J, Nadiejda E, Robles R, Del Aguila JM, Cunha P, Vassilenko V, Rodilla E, Sanchez Munoz-Torrero JF. Automated Office Blood Pressure Measurements in Waiting Room or Isolated Room for Diagnosis and Phenotyping of Hypertension. J Am Heart Assoc. 2025 Oct 21;14(20):e038011. doi: 10.1161/JAHA.124.038011. Epub 2025 Oct 14. PMID 41085208